CLINICAL TRIAL: NCT01389063
Title: Maraviroc Abacavir STudy - Effect on Endothelial Recovery
Acronym: MASTER
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: S.F.L. van Lelyveld (Other)
Responsible Party: Sponsor-Investigator, S.F.L. van Lelyveld, Coordinating investigator, UMC Utrecht
Organization: UMC Utrecht (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MASTER2010
Record Dates: First submitted 2011-07-05; First posted 2011-07-07 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-12

CONDITIONS: Endothelial Dysfunction
Keywords: endothelial function; CCR5 receptor; Maraviroc; Abacavir; Flow Mediated Dilatation; EndoPAT
MeSH Terms: conditions — Diabetes Mellitus, Insulin-Dependent, 22 | interventions — Maraviroc

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Active Comparator): HAART of subjects in arm A will be intensified with maraviroc during week 1-8.
  Interventions: Drug: Maraviroc
- Arm B (Active Comparator): HAART of subjects enrolled in arm B will be intensified with maraviroc during week 9-16
  Interventions: Drug: Maraviroc

INTERVENTIONS:
Drug: Maraviroc — HAART of subjects enrolled in arm A will be intensified with maraviroc during week 1-8.
  Other Names: Celsentri

SUMMARY:
HIV infected patients treated with abacavir might have a higher risk for the occurrence of cardiovascular events. At time of writing of this protocol the underlying mechanism is not yet elucidated, however some studies find impaired endothelial function and elevated markers of chronic inflammation in these patients,suggesting a higher lever of chronic inflammation. Recently maraviroc (Celsentri®), a CCR5-receptor antagonist, became available for treatment of patients infected with HIV-1.

Improvement of endothelial function may be a potential beneficial side effect of treatment with maraviroc, due to the potential reduction of immune activation and chronic inflammation as a result of blocking the CCR5-coreceptor. Moreover, treatment intensification of HAART with maraviroc in patients with suppressed plasma HIV_RNA may decrease plasma HIVRNA below the cut-off of 50 copies/ml as well.

The investigators hypothesize that maraviroc intensification therapy in patients on an abacavir-containing regimen will improve endothelial function.

The objectives of this study are: First, to assess the effect of addition of maraviroc to an abacavir-containing regimen on endothelial function; second, to assess the effect of this intervention on markers of immune activation and chronic inflammation, and on plasma HIV-RNA below 50 copies/ml.

DETAILED DESCRIPTION:
The MASTER study is a phase IV, randomized, open label, cross-over, intervention study. Study subjects who are on stable abacavir-containing regimen will be randomized into two arms. In arm A maraviroc will be added to their regimen at baseline, while study subjects in arm B will continue their abacavir-containing regimen. After 8 weeks, cross-over of the study arms will be performed. Subjects in arm A will then stop maraviroc, while in subjects in arm B maraviroc will be added to their regimen (for 8 weeks again). The total duration of the study will be 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* HIV-1 infection
* Treatment with antiretroviral regimen containing abacavir for at least the previous 3 months
* Undetectable plasma HIV RNA (50 cp/ml) for at least 6 months (one 'blip' allowed, which is defined as a detectable plasma HIV-RNA level between 50 and 400 copies/ml, preceded and followed by undetectable (<50 copies/ml) plasma HIV-RNA measurements)
* CD4+ cell count > 200 cells/μL
* Signed informed consent

Exclusion Criteria:

* Pregnancy
* Breastfeeding
* Allergy for peanuts or soya
* Hypersensitivity for maraviroc
* Treatment of underlying malignancy
* Acute infection in the preceding 30 days
* Renal insufficiency requiring hemodialysis
* Acute or decompensated chronic hepatitis
* Modification of antiretroviral regimen in the previous 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-09 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Change in flow-mediated dilatation (FMD) of the brachial artery after 8 weeks of maraviroc treatment as compared to the control group | After 8 weeks of treatment (cross-over)

SECONDARY OUTCOMES:
Change in markers of chronic inflammation | Baseline, week 2, week 4, week 8, week 10, week 12 and week 16
Change in markers of immune activation | Baseline, week 2, week 4, week 8, week 10, week 12 and week 16
Change in markers of endothelial function | Baseline, week 2, week 4, week 8, week 10, week 12 and week 16
Changes in plasma HIV-RNA below 50 copies/ml | Baseline, week 8, week 16
Change in endothelial function measured by EndoPAT | baseline, week 8, week 16

CONTACTS AND LOCATIONS:
Overall Officials: A IM Hoepelman, MD, PhD, Principal Investigator — UMC Utrecht
Locations (1):
- University Medical Center Utrecht, Utrecht, Netherlands

REFERENCES:
- [Derived] Krikke M, Tesselaar K, Arends JE, Drylewicz J, Otto SA, van Lelyveld SF, Visseren FJ, Hoepelman AI. Maraviroc Intensification Improves Endothelial Function in Abacavir-Treated Patients, an Open-Label Randomized Cross-Over Pilot Study. Infect Dis Ther. 2016 Sep;5(3):389-404. doi: 10.1007/s40121-016-0115-0. Epub 2016 Jun 14. PMID 27300170